CLINICAL TRIAL: NCT04287907
Title: The Utility of Qualitative End Tidal CO2 Detector in Providing Effective Ventilation During Resuscitation of Preterm Newborns: A Pilot Randomized Controlled Trial
Brief Title: Use of CO2 Detectors to Help Provide Effective Breaths During Resuscitation of Preterm Newborns
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: KK Women's and Children's Hospital (Other Government)
Responsible Party: Principal Investigator, Kong Juin Yee, Consultant Neonatologist, KK Women's and Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2016/2405
Record Dates: First submitted 2020-02-19; First posted 2020-02-27 (Actual); Last update posted 2023-10-04 (Actual); Status verified 2023-10

CONDITIONS: Preterm Birth
Keywords: end tidal carbon dioxide; mask ventilation; neonatal resuscitation
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Monitor (Experimental): Qualitative End Tidal Co2 detector will be attached to the face mask used to provide mask ventilation to the preterm baby before connected to the T piece resuscitator. Respiratory function monitor sensor will be placed within circuit to measure parameters e.g. PIP, PEEP, FiO2, tidal volume.
  Interventions: Device: Monitor Group
- Control (No Intervention): face mask used to provide mask ventilation to the preterm baby will be connected directly to the T piece resuscitator. Respiratory function monitor sensor will be placed within circuit to measure parameters e.g. PIP, PEEP, FiO2, tidal volume.

INTERVENTIONS:
Device: Monitor Group — Use of colorimetric end tidal CO2 to guide provider during provision of mask ventilation, where colour change indicates effective breaths
  Arms: Monitor

SUMMARY:
Effective ventilation is the single most vital intervention to improve outcome of resuscitation in the neonatal population. Assessments of effective ventilations are based on clinical parameters, but may be difficult due to inexperienced personnel as well as observer variability. End tidal CO2 detectors (ETCO2) have been shown to improve effective ventilation in manikin model as well as in video recordings of selective infants where obstructive breaths were recognized objectively by means of lack of colour change.

This is a trial evaluating the use of a qualitative end tidal CO2 monitor device during mask ventilation in the delivery room. The investigators hypothesize that using a colorimetric carbon dioxide detector during mask ventilation, it could facilitate recognition of obstructed breaths and reduce the duration of bradycardia and desaturations.

ELIGIBILITY:
Inclusion Criteria:

Preterm infants 24+0/7 to 32+0/7 weeks who require mask ventilation during resuscitation

Exclusion Criteria:

1. Infants with impaired pulmonary circulation (eg. Cardiac arrest, pulmonary atresia, severe pulmonary stenosis
2. Infants with congenital airway anomalies

Max Age: 60 Minutes | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 50 (Actual)
Dates: Start 2019-06-06 (Actual); Primary Completion 2021-04-10 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Bradycardia and Desaturation Duration | This outcome will be obtained immediately after birth when available on pulse oximetry
  Duration of bradycardia (HR<100beats per minute) + Desaturation (SpO2 readings below recommended target during respective minutes of life after birth

SECONDARY OUTCOMES:
Delivery room intubation | During resuscitation course at birth
  This outcome will be counted as yes if infant required endotracheal intubation in the delivery room
Delivery room chest compressions | During resuscitation course at birth
  This outcome will be counted as yes if infant required chest compressions in the delivery room
Delivery room peak inspiratory pressure (PIP) | During resuscitation course at birth
  Peak inspiratory pressure (PIP) used during mask ventilation during resuscitation after birth, measured as cmH20
Delivery room positive end expiratory pressure (PEEP) | During resuscitation course at birth
  Positive end expiratory pressure (PEEP) used during mask ventilation during resuscitation after birth, measured as cmH20
Delivery room fraction of inspired oxygen level (FiO2) | During resuscitation course at birth
  Fraction of inspired oxygen level (FiO2) measured using an oxygen analyser within the ventilating circuit during mask ventilation (ranges from 0.21-1.0)
Tidal volume during resuscitation | During resuscitation course at birth
  Tidal volume (ml/kg) measured using a respiratory function monitor sensor attached to the mask during mask ventilation
Mask leakage during resuscitation | During resuscitation course at birth
  mask leakage (%) measured and calculated using a respiratory function monitor during mask ventilation
Apgar Scores | During resuscitation course at birth
  Apgar score with a scale of 0-10 (0 being the worst and 10 the best) obtained by adding points for heart rate, respiratory effort, muscle tone, reflex, and colour to represent the condition of newborn baby after birth. Scores are assigned at at 1 and 5 minutes of life respectively, with extension after 10 minutes if initial scores are low
Admission blood gas partial pressure of carbon dioxide (pCO2) levels | During inpatient hospital course, usually 2-3 months
  first blood gas pCO2 levels in mmHg
Occurrence of air leak syndromes | During inpatient hospital course, usually 2-3 months
  pneumothorax, pneumomediastinum confirmed on x ray
Duration of assisted ventilation before discharge | During inpatient hospital course, usually 2-3 months
  ventilation days on mechanical ventilator or continuous positive airway pressure (CPAP) respectively
incidence of severe intraventricular hemorrhage (IVH) | During inpatient hospital course, usually 2-3 months
  ultrasound finding of grade3-4 intraventricular hemorrhage
incidence of necrotizing enterocolitis (NEC) | During inpatient hospital course, usually 2-3 months
  diagnosis of NEC proven by abdominal X-rays, classified as Bell Stage II
incidence of chronic lung disease (CLD) | During inpatient hospital course, usually 2-3 months
  diagnosed when there is a need for oxygen at 36 weeks post menstrual age
incidence of severe retinopathy of prematurity (ROP) | During inpatient hospital course, usually 2-3 months
  diagnosed when there is a need for laser surgery for treatment of ROP

OTHER OUTCOMES:
Number of corrective measures performed | During resuscitation at birth
  Number of corrective measures performed to overcome ineffective mask ventilation observed on video recording of resuscitation

CONTACTS AND LOCATIONS:
Overall Officials: Juin Yee Kong, MD, Principal Investigator — KK Women's and Children's Hospital
Locations (1):
- KK Women's and Children's Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Finer NN, Rich W, Wang C, Leone T. Airway obstruction during mask ventilation of very low birth weight infants during neonatal resuscitation. Pediatrics. 2009 Mar;123(3):865-9. doi: 10.1542/peds.2008-0560. PMID 19255015
- [Background] Leone TA, Lange A, Rich W, Finer NN. Disposable colorimetric carbon dioxide detector use as an indicator of a patent airway during noninvasive mask ventilation. Pediatrics. 2006 Jul;118(1):e202-4. doi: 10.1542/peds.2005-2493. Epub 2006 Jun 26. PMID 16801392
- [Background] Hawkes GA, Finn D, Kenosi M, Livingstone V, O'Toole JM, Boylan GB, O'Halloran KD, Ryan AC, Dempsey EM. A Randomized Controlled Trial of End-Tidal Carbon Dioxide Detection of Preterm Infants in the Delivery Room. J Pediatr. 2017 Mar;182:74-78.e2. doi: 10.1016/j.jpeds.2016.11.006. Epub 2016 Dec 9. PMID 27939108
- [Derived] Kong JY, Quek BH, Lim CSE, Sultana R, Ng YYV, Rajadurai VS, Yeo KT. Colorimetric CO2 Detector to Improve Effective Mask Ventilations in Very Preterm Infants: A Pilot Randomized Controlled Study. Neonatology. 2024;121(4):494-502. doi: 10.1159/000538083. Epub 2024 Mar 27. PMID 38537615